CLINICAL TRIAL: NCT03585868
Title: Evaluation of the Effects of a COcoa Supplement to Reduce FRailty in the Elderly: COFRE a Randomized Clinical Trial
Brief Title: Effects of COcoa Supplement in FRail Elderly Subjects (COFRE)
Acronym: COFRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Polytechnic Institute, Mexico (Other)
Responsible Party: Principal Investigator, Guillermo Ceballos Reyes, Professor, National Polytechnic Institute, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COFRE-LIICM
Record Dates: First submitted 2018-05-16; First posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Sarcopenia; Frail Elderly Syndrome
Keywords: flavonoids
MeSH Terms: conditions — Sarcopenia | interventions — Flavonoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Beverage without flavonoids
  Interventions: Other: Placebo
- No Flavonoids (Sham Comparator): Beverage with alkalinized cocoa which eliminates flavonoid content
  Interventions: Dietary Supplement: No Flavonoids
- Flavonoids (Experimental): Beverage with a flavonoid rich mixture
  Interventions: Other: Flavonoids

INTERVENTIONS:
Other: Placebo — Beverage with no flavonoids
  Arms: Placebo
Other: Flavonoids — Flavonoids-enriched cacao beverage
  Arms: Flavonoids
Dietary Supplement: No Flavonoids — Beverage with alkalinized cocoa which eliminates flavonoid content
  Arms: No Flavonoids

SUMMARY:
The study use a double blind, placebo-controlled design enrolling male and female subjects between 55-90 yo to evaluate the effect of daily consumption of a cocoa beverage on anthropometric, metabolic, oxidative stress, physical performance and quality of life.

DETAILED DESCRIPTION:
The study use a double blind, placebo-controlled design enrolling male and female subjects between 55-90 yo randomly assigned to consumption of a flavonoid rich mixture (flavonoids; F), alkalinized cocoa which eliminates flavonoid content (no flavonoids; NF) or placebo. All beverages had similar physical characteristics and flavor. Cocoa beverages were provided in individual sachets containing a dry powder that was reconstituted with water just before consumption. Subjects were instructed as above to maintain their usual lifestyle, to limit intake of high caloric foods and flavonoid-containing foods and beverages, and to walk for 30 min/day.

To determine the effect of flavonoids, study evaluates anthropometric measures, metabolic parameters as glycemia and a lipid profile (triglycerides, total cholesterol, high-density lipoprotein cholesterol and low-density lipoprotein cholesterol). To evaluate oxidative stress damage as lipid oxidation is measured with the malondialdehyde (MDA) assay. Protein carbonylation is measured using an assay for detection of carbonyl groups that relies on 2,4-dinitrophenylhydrazine (DNPH) as a substrate. The investigators also evaluate interleukin-6 and tumor necrosis factor levels.

For physical performance is evaluated the handgrip strength, and mobility assesment with the following test: Six-minute walk test, two-minute step, sit-up test and the up & go test.

The investigators also assessed quality of life using the Health Related QoL (EQ-5D) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Sex: both
* Age: 55-90 yo
* Waist circumference: Women > 80 cm, Men > 90 cm
* HDL-c: Women < 50 mg/dL, Men < 40 mg/dL
* Triglycerides: ≥ 150 mg/dL
* Glycemia: ≈100 mg/dL
* Hand strength: Women< 20 kg, Men < 30 kg
* Up & Go test: > 10 seconds

Non-inclusion criteria:

* Any active infections
* Malignancies
* Habitual consumers of antioxidant supplements and cocoa products
* Use of benzodiazepines or protein supplements

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Blood glucose | At 90 days
  Fasting blood level
Serum triacylglycerol concentration | At 90 days
  Fasting blood level
Serum total cholesterol | At 90 days
  Fasting blood level
Serum HDL cholesterol | At 90 days
  Fasting blood level
Serum LDL cholesterol | At 90 days
  Fasting blood level
Lipid oxidation | At 90 days
  Serum malondialdehyde Levels
Protein oxidation | At 90days
  Serum protein carbonylation Levels

SECONDARY OUTCOMES:
Handgrip strength | At 60 days
  Measures static force in kilograms that the hand can squeeze around a dynamometer
Up and go test | At 60 days
  Measures time in seconds, a subject can rise and walk a 3-meter line and return to sit down
Six-minute walk test | 6 minutes
  Measures maximum distance in meters, a subject can walk at their normal gait and pace during 6 minutes
Two-minute step in place test | 2 minutes
  Measures number of times a subject can rise each knee to the hip level during 2 minutes.
Sit-up test | 30 seconds
  Measures number of times a subject can rise and sit-down in place during 30 seconds
EQ-5D questionnaire | At 60 days
  Self-administered health index that explores five domains
Analog Visual Scale | At 60 days
  Use of a Analog Visual Scale to measure the quality of life, graded 0 (worst) to 100 (best) for the perception of wellbeing.

REFERENCES:
- [Derived] Munguia L, Rubio-Gayosso I, Ramirez-Sanchez I, Ortiz A, Hidalgo I, Gonzalez C, Meaney E, Villarreal F, Najera N, Ceballos G. High Flavonoid Cocoa Supplement Ameliorates Plasma Oxidative Stress and Inflammation Levels While Improving Mobility and Quality of Life in Older Subjects: A Double-Blind Randomized Clinical Trial. J Gerontol A Biol Sci Med Sci. 2019 Sep 15;74(10):1620-1627. doi: 10.1093/gerona/glz107. PMID 31056655